CLINICAL TRIAL: NCT02194049
Title: Phase I Trial of Cisplatin and Etoposide Plus BKM120 in Advanced Solid Tumors, With an Emphasis on Small Cell Lung Cancer
Brief Title: Cisplatin, Etoposide and PI3K Inhibitor BKM120 in Treating Patients With Advanced Solid Tumors or Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#239; 470970 (Registry Identifier: UC Davis); CBKM120ZUS38T (Other: Novartis); UCDCC#239 (Other: University of California at Davis Cancer Center); NCI-2014-00218 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-07-10; First posted 2014-07-18 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2016-06

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — NVP-BKM120; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM 120, cisplatin, etoposide (Experimental): Patients receive PI3K Inhibitor BKM120 PO QD on days 1-21, cisplatin IV over 2 hours on day 1 and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BKM120; Drug: cisplatin; Drug: etoposide

INTERVENTIONS:
Drug: BKM120 — Given PO
  Other Names: PI3K_Inhibitor_BKM120
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213

SUMMARY:
This phase I trial studies the side effects and the best dose of PI3K inhibitor BKM120 when given together with cisplatin and etoposide in treating patients with advanced solid tumors or small cell lung cancer. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing , or by stopping them from spreading. PI3K inhibitor BKM120 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving PI3K inhibitor BKM120 with cisplatin and etoposide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of combining BKM120 (PI3K inhibitor BKM120) with cisplatin and etoposide in advanced solid tumors, with emphasis on small cell lung cancer (SCLC).

SECONDARY OBJECTIVE:

I. To determine the MTD (maximally tolerated dose) of BKM120 in combination with cisplatin/etoposide.

II. To describe the dose limiting toxicities (DLT) and toxicity profile associated with BKM120 in combination with cisplatin/etoposide.

III. To determine the preliminary efficacy of BKM120 in combination with cisplatin/etoposide in an expanded cohort of patients with SCLC.

IV. To characterize the pharmacokinetic (PK) parameters of BKM120 in this combination.

V. To collect blood samples for future exploratory biomarker analysis.

OUTLINE: This is a dose-escalation study of PI3K inhibitor BKM120.

Patients receive PI3K Inhibitor BKM120 orally (PO) once daily (QD) on days 1-21, cisplatin intravenously (IV) over 2 hours on day 1 and etoposide IV over 1 hour on days 1-3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of treatment, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proven advanced solid tumors
* =< 3 chemotherapy regimens for metastatic disease; any number of prior targeted or biologic therapies is allowed; (in the expansion cohort, patients must be chemo naïve)
* ECOG performance status =< 2
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hb) > 9 g/dL
* Total calcium (corrected for serum albumin) within normal limits (bisphosphonate use for malignant hypercalcemia control is not allowed)
* Magnesium >= the lower limit of normal
* Potassium within normal limits for the institution
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range (or =< 3.0 x upper limit of normal (ULN) if liver metastases are present)
* Serum bilirubin within normal range (or =< 1.5 x ULN if liver metastases are present; or total bilirubin =< 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
* Serum creatinine =< 1.5 x ULN or calculated clearance >= 60 mL/min
* Serum albumin >= 3 g/dl
* Serum amylase =< ULN
* Serum lipase =< ULN
* Fasting plasma glucose =< 120 mg/dL (6.7 mmol/L)
* International normalized ratio (INR) =< 2
* Ability to swallow pills
* Negative serum pregnancy test

Exclusion Criteria:

* Received prior treatment with a P13K inhibitor
* Received > 300 mg/m^2 of cisplatin and/or for whom cisplatin would not be beneficial
* Prior treatment with any investigational drug within the preceding 3 weeks
* Known hypersensitivity to BKM120 or to its excipients
* Untreated brain metastases are excluded
* Acute or chronic liver, renal disease or pancreatitis
* Following mood disorders as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire
* Diarrhea >= CTCAE grade 2
* Active cardiac disease
* History of cardiac dysfunction
* Poorly controlled diabetes mellitus or steroid-induced diabetes mellitus
* Other concurrent severe and/or uncontrolled concomitant medical conditions
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection); patients with unresolved diarrhea will be excluded as previously indicated
* Treated with any hematopoietic colony-stimulating growth factors
* Currently receiving treatment with medication with a known risk to prolong the QT interval or inducing torsades de pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
* Chronic treatment with steroids or another immunosuppressive agent
* Herbal medications and certain fruits within 7 days prior to starting study drug
* Treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Intravenous chemotherapy or targeted anticancer therapy =< 4 weeks
* Any continuous or intermittent oral small molecule therapeutics
* Received wide field radiotherapy =< 4 weeks or limited field radiation for palliation =< 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Undergone major surgery =< 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Currently taking therapeutic doses of warfarin sodium or any other Coumadin-derivative anticoagulant
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control
* Known diagnosis of HIV infection
* History of another active malignancy
* Unable or unwilling to abide by the study protocol or cooperate fully with the investigator treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events of combining daily BKM120 with cisplatin and etoposide as graded by the National Cancer Institute (NC) CTCAE version 4.0 | Up to 28 days post-treatment
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity, time of onset (i.e. course number), duration, and reversibility or outcome.

SECONDARY OUTCOMES:
MTD defined as the highest dose tested in which fewer than 33% of patients experience DLT attributed to the study drugs when at least 6 patients were treated at that dose, as graded by NCI CTCAE version 4.0 | 21 days
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity, time of onset (i.e. course number), duration, and reversibility or outcome.
Response rate assessed by computed tomography (CT) scan based on Response Evaluation Criteria In Solid Tumors (RECIST) | Up to 30 days
  Response rate among patients with measurable disease will be summarized by exact binomial confidence intervals
Overall survival | Up to 30 days
  Survival will be summarized with Kaplan-Meier plots to describe the outcome of patients treated on this protocol. Median survival time will be estimated using standard life table methods.
Time to progression (TTP) based on RECIST | Up to 30 days
  TTP will be summarized with Kaplan-Meier plots to describe the outcome of patients treated on this protocol. Median time to progression will be estimated using standard life table methods.
Pharmacokinetic analysis | Baseline, at 1, 2, 4, 6, and 24 hours of day 1 of course 1, baseline day 15 of course 1, and at 1 and 2 hours post-dose on day 1 of course 2
  Pharmacokinetic analysis will use non-linear curve fitting methods to estimate the mean peak concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kelly, Principal Investigator — University of California, Davis
Locations (1):
- University of California at Davis Cancer Center, Sacramento, California, United States